CLINICAL TRIAL: NCT03018132
Title: The PROVIDE Study; Preeclampsia Research on Vitamin D, Inflammation, & Depression
Brief Title: Preeclampsia Research on Vitamin D, Inflammation, & Depression
Acronym: PROVIDE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Maternal Mental Health NOW (Unknown)
Responsible Party: Principal Investigator, Eynav Accortt, Assistant Professor, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pro00044664
Record Dates: First submitted 2016-12-08; First posted 2017-01-11 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Pre-Eclampsia; Depression; Inflammation; Vitamin D Deficiency
Keywords: perinatal mental health
MeSH Terms: conditions — Pre-Eclampsia; Depression; Inflammation; Vitamin D Deficiency | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mental Health Screening Education and Referral (Other): Investigators will prospectively assign all 200 women to this screening, education and referral intervention, without concurrent comparison or control groups, to study the cause-and-effect relationship between a health-related intervention and a health outcome. The health-related intervention, in this case, is an educational program and related process-of-care changes.
  Interventions: Other: mental health screening, education and referral program

INTERVENTIONS:
Other: mental health screening, education and referral program — I. Psychosocial assessments:
  1. Mental health screening for: (1) depressive symptoms with the EPDS, (2) post-traumatic stress symptoms with the IES, (3) for perceived stress with the PSS (4) for anxiety with the OASIS.
  2. Exercise, smoking & substance use, sleep and nutrition.
  II. If women are above cutoff values the SCID will be conducted.
  III. Education and referral information via Maternal Mental Health NOW:
  1. All receive a brochure entitled, Speak Up When You Are Down
  2. If above cutoffs, participants will also receive referral information; and will be scheduled for a SCID
  3. Trained study staff will review the brochure and show the woman how to use the MMHN online referral system to input their zip code and find preferred maternal mental health practitioners.
  IV. Follow up with a survey at 3 months postpartum: acceptability of screening, benefit of referral service, and outcome of this referral.

SUMMARY:
This study is designed to comprehensively investigate the anti-inflammatory role of vitamin D in reproductive aged women, and its association with preeclampsia and depression. Findings will have substantial impact providing new information implicated in the development of preeclampsia (a condition that may include hypertension, tissue swelling caused by excessive fluid, and kidney stress) and postpartum depression (after birth).

Additionally, the study is designed to understand how early mental health screening and evaluation can help pregnant women reduce their risk of developing postpartum depression. Testing the acceptability and effectiveness of this mental health screening, education and referral program at Cedars-Sinai Medical Center will provide valuable patient centered qualitative and quantitative data that can be used in future services planning.

The study will enroll up to 200 pregnant women (in third trimester of pregnancy) in total.

DETAILED DESCRIPTION:
Background information

The PROVIDE study tests the hypothesis that low vitamin D levels and increased inflammatory activity in pregnant women contributes to increased risk of preeclampsia and postpartum depression (PPD). Preeclampsia is a multisystem disorder of pregnancy commonly characterized by hypertension that occurs after 20 weeks of gestation in a woman with previously normal blood pressure accompanied by proteinuria. One pathway thought to lead to preeclampsia is chronic subclinical inflammation. Likewise, inflammation is elevated in women with major depressive disorder (MDD) and PPD and may therefore be a common physiological pathway connecting depression with preeclampsia. In addition, vitamin D deficiency, which is common in pregnancy and the postpartum period is associated with depressive symptomatology, prenatal inflammation and adverse birth outcomes, particularly preeclampsia. Research has shown that vitamin D acts as an anti-inflammatory agent regulating placental function to promote tolerance of the fetus. Prior work demonstrated that among women with elevated prenatal inflammation, higher prenatal vitamin D status was associated with lower PPD symptoms. This research tests the hypothesis that vitamin D deficiency places women with higher levels of inflammatory cytokines at highest risk for preeclampsia and PPD. Findings will have substantial impact providing new information about inflammatory mechanisms implicated in the development of preeclampsia and PPD, and will support future research, such as vitamin D supplementation to reduce risk for preeclampsia and depression.

The study also seeks a better understanding of several important biopsychosocial consequences of developing preeclampsia. In pregnancy, 8-13% of women are diagnosed with MDD, which can lead to postpartum depression (PPD) and adverse birth outcomes, specifically low birth weight and preeclampsia. Although maternal depression is associated with negative consequences for the mother, her infant and family, low rates of diagnosis and treatment for perinatal depression are common in medical settings. Rapid diagnosis and treatment is essential because the episodes are lengthy and psychosocial symptoms (including anxiety) increase with the duration of the disorder. Screening is important because it is the first step in the pathway to treatment. This study tests the acceptability and benefits of a mental health screening, education and referral program in women with and without preeclampsia. With assistance from a community partner, Maternal Mental Health-NOW (formerly the L.A. County Perinatal Mental Health Task Force), findings will provide valuable patient centered qualitative and quantitative data that can be used in future services planning. This is timely work. In 2015 ACOG recommended that clinicians screen patients at least once during the perinatal period for depression and anxiety symptoms. Post-traumatic stress symptoms are particularly common after experiencing an adverse pregnancy outcome, and approximately 9% develop Post-traumatic stress disorder (PTSD). Increased risk of major depression (40-50%) comorbid with PTSD can lead to decreased maternal bonding with infant and other long term adverse mental and physical health repercussions for the mother, child and family. Screening therefore must be coupled with appropriate follow-up and treatment when indicated, and systems should be in place to ensure follow-up for diagnosis and treatment. Most recently (2016), the US Preventive Services Task Force (USPSTF) made perinatal depression screening recommendations, adding that data are lacking on both the accuracy of screening and the benefits and harms of treatment in pregnant women. The authors highlight that research is needed to assess barriers to establishing adequate systems of care and how these barriers can be addressed.

Very little is known from the patient perspective regarding acceptance and benefits of mental health screening. There is even less understanding of the variation in preferences and need for these services in women who experience preeclampsia, for whom PPD rates are even higher. The perinatal period is an opportune time for screening and mental health education due to the frequency of contact with health care providers, unfortunately rates of diagnosis and treatment for perinatal depression are low in medical settings. New parents are often highly motivated to seek help in effecting change for the sake of their offspring and potential reduction in intergenerational family dysfunction. The perinatal period thus provides clinicians with a unique opportunity to consider universal psychosocial assessment as part of mainstream maternity and postnatal care. Early identification and treatment of psychosocial morbidity are especially important in relation to the functioning of the family unit and the critical parent-infant relationship with potential to positively impact on the health of the next generation. Routine depression screening and referral has been supported by RCTs in Primary Care. RCT work has not been conducted in the perinatal period or in the OB/GYN setting, however screening, education, and referral programs in obstetric settings have been well accepted by patients. Overall, mental health care might be most acceptable if provided as part of routine obstetrical care. Mental health screening and treatment might also be more beneficial in the subset of women who experience adverse pregnancy complications. Results from this mental health screening program will allow for early identification and intervention at a time when women are at highest risk for mental health complications, after an adverse complication such as preeclampsia.

Objectives and purpose

To our knowledge, no studies have comprehensively investigated the anti-inflammatory role of vitamin D in depressed reproductive aged women, and its association with adverse pregnancy outcomes. Findings will have substantial impact providing new information about inflammatory mechanisms implicated in the development of preeclampsia and PPD, and will support future intervention research, including vitamin D supplementation, focused on alleviating these effects. Additionally, testing the acceptability and effectiveness of a new mental health screening, education and referral program at Cedars-Sinai Medical Center (CSMC) will provide valuable patient centered qualitative and quantitative data that can be used in future services planning.

PROVIDE study hypotheses will be tested in a new cohort (N=200) recruited in the third trimester from CSMC Childbirth and Education classes, the Prenatal Diagnostic Center (PDC), or in the Maternal-Fetal Care Unit (MFCU, for those diagnosed with Preeclampsia); and followed through delivery and 2 time points (4 weeks and 3 months) postpartum. A targeted sampling strategy over a two-year period will result in 100 women who experience preeclampsia and 100 women who do not.

Specific Aim 1: Determine to what extent prenatal vitamin D deficiency (defined clinically as serum 25(OH)D < 20 ng/ml48) will be associated with increases in prenatal inflammatory cytokines (e.g. hs-CRP and Interleukin-6), prenatal depressive symptoms, and preeclampsia.

Hypothesis: Women who experience lower prenatal vitamin D levels will exhibit an increased likelihood of experiencing prenatal depression, preeclampsia, and postpartum depression. These effects will be greatest in those with high levels of prenatal inflammatory cytokines.

Specific Aim 2: Determine to what extent women who have preeclampsia will have increases in postpartum inflammatory cytokines, vitamin D deficiency and PPD.

Hypothesis: Compared to those who do not experience preeclampsia, women with preeclampsia will have higher postpartum levels of inflammatory cytokines, lower postpartum vitamin D levels, and increased symptoms of PPD.

Specific Aim 3: Determine to what extent a mental health program that includes screening, education and referral is acceptable to pregnant women and effective in reducing symptoms of postpartum depression, anxiety and/or stress following preeclampsia.

Hypothesis: Women in the preeclampsia + depression group will rate the mental health program as more acceptable and beneficial, and will follow up on referral suggestions more than depressed-only group.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Minimum 18 years of age
* Patient at Cedars Sinai Medical Center, Los Angeles, CA
* Between 20 and 40 weeks gestation (majority recruited at start of 3rd trimester between 26-32 weeks)
* English or Spanish language preference

Exclusion Criteria:

* Any diagnosis of psychosis, past or current (evident by either meds taken via medical intake, or in clinical assessment - SCID)
* Current substance abuse (evident either via medical intake, or in clinical assessment - SCID)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | 5 months
  as measured by reliable and validated screening tool (EPDS)
Depression Diagnosis | 5 months
  as measured by diagnostic interview (SCID)

SECONDARY OUTCOMES:
Anxiety symptoms | 5 months
  as measured by the OASIS
Post-traumatic stress symptoms | 5 months
  as measured by the IES
Perceived stress | 5 months
  as measured by the PSS
Acceptability of Mental Health Program | 5 months
  Results will be based on data from structured (Likert-scale) surveys completed at 4 time points, from the patient perspective
Benefits of Mental Health Program | 5 months
  Results will be based on data from the follow-up structured (Likert-scale) survey
Feasibility of Mental Health Program | 5 months
  The program's feasibility and MMH-Now training will be rated by clinic staff according to structured surveys completed at multiple time points, e.g. pre/post training.
Inflammation_IL6 | 5 months
  as measured by serum Interleukin-6
Inflammation_CRP | 5 months
  as measured by serum hs_CRP
Vitamin D deficiency | 5 months
  as measured by serum 25(OH)D levels

CONTACTS AND LOCATIONS:
Overall Officials: Eynav Accortt, PhD, Principal Investigator — Cedars Sinai Medical Center Department of OBGYN
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller DA. Hypertension in pregnancy. Diagnosis and treatment obstetrics and gynecology 2003;10:318.
- [Background] Christian LM. Psychoneuroimmunology in pregnancy: immune pathways linking stress with maternal health, adverse birth outcomes, and fetal development. Neurosci Biobehav Rev. 2012 Jan;36(1):350-61. doi: 10.1016/j.neubiorev.2011.07.005. Epub 2011 Jul 19. PMID 21787802
- [Background] Xiao JP, Yin YX, Gao YF, Lau S, Shen F, Zhao M, Chen Q. The increased maternal serum levels of IL-6 are associated with the severity and onset of preeclampsia. Cytokine. 2012 Dec;60(3):856-60. doi: 10.1016/j.cyto.2012.07.039. Epub 2012 Aug 22. PMID 22921280
- [Background] Pinheiro MB, Martins-Filho OA, Mota AP, Alpoim PN, Godoi LC, Silveira AC, Teixeira-Carvalho A, Gomes KB, Dusse LM. Severe preeclampsia goes along with a cytokine network disturbance towards a systemic inflammatory state. Cytokine. 2013 Apr;62(1):165-73. doi: 10.1016/j.cyto.2013.02.027. Epub 2013 Mar 21. PMID 23523008
- [Background] Dantzer R, O'Connor JC, Freund GG, Johnson RW, Kelley KW. From inflammation to sickness and depression: when the immune system subjugates the brain. Nat Rev Neurosci. 2008 Jan;9(1):46-56. doi: 10.1038/nrn2297. PMID 18073775
- [Background] Howren MB, Lamkin DM, Suls J. Associations of depression with C-reactive protein, IL-1, and IL-6: a meta-analysis. Psychosom Med. 2009 Feb;71(2):171-86. doi: 10.1097/PSY.0b013e3181907c1b. Epub 2009 Feb 2. PMID 19188531
- [Background] Miller AH, Maletic V, Raison CL. Inflammation and its discontents: the role of cytokines in the pathophysiology of major depression. Biol Psychiatry. 2009 May 1;65(9):732-41. doi: 10.1016/j.biopsych.2008.11.029. Epub 2009 Jan 15. PMID 19150053
- [Background] Osborne LM, Monk C. Perinatal depression--the fourth inflammatory morbidity of pregnancy?: Theory and literature review. Psychoneuroendocrinology. 2013 Oct;38(10):1929-52. doi: 10.1016/j.psyneuen.2013.03.019. Epub 2013 Apr 20. PMID 23608136
- [Background] Christian LM, Franco A, Glaser R, Iams JD. Depressive symptoms are associated with elevated serum proinflammatory cytokines among pregnant women. Brain Behav Immun. 2009 Aug;23(6):750-4. doi: 10.1016/j.bbi.2009.02.012. Epub 2009 Mar 1. PMID 19258033
- [Background] Ginde AA, Sullivan AF, Mansbach JM, Camargo CA Jr. Vitamin D insufficiency in pregnant and nonpregnant women of childbearing age in the United States. Am J Obstet Gynecol. 2010 May;202(5):436.e1-8. doi: 10.1016/j.ajog.2009.11.036. Epub 2010 Jan 12. PMID 20060512
- [Background] Murphy PK, Mueller M, Hulsey TC, Ebeling MD, Wagner CL. An exploratory study of postpartum depression and vitamin d. J Am Psychiatr Nurses Assoc. 2010 May;16(3):170-7. doi: 10.1177/1078390310370476. PMID 21659271
- [Background] Fu CW, Liu JT, Tu WJ, Yang JQ, Cao Y. Association between serum 25-hydroxyvitamin D levels measured 24 hours after delivery and postpartum depression. BJOG. 2015 Nov;122(12):1688-94. doi: 10.1111/1471-0528.13111. Epub 2014 Sep 19. PMID 25233808
- [Background] Anglin RE, Samaan Z, Walter SD, McDonald SD. Vitamin D deficiency and depression in adults: systematic review and meta-analysis. Br J Psychiatry. 2013 Feb;202:100-7. doi: 10.1192/bjp.bp.111.106666. PMID 23377209
- [Background] Cassidy-Bushrow AE, Peters RM, Johnson DA, Li J, Rao DS. Vitamin D nutritional status and antenatal depressive symptoms in African American women. J Womens Health (Larchmt). 2012 Nov;21(11):1189-95. doi: 10.1089/jwh.2012.3528. Epub 2012 Jul 23. PMID 22823176
- [Background] Hoogendijk WJ, Lips P, Dik MG, Deeg DJ, Beekman AT, Penninx BW. Depression is associated with decreased 25-hydroxyvitamin D and increased parathyroid hormone levels in older adults. Arch Gen Psychiatry. 2008 May;65(5):508-12. doi: 10.1001/archpsyc.65.5.508. PMID 18458202
- [Background] Bobbitt KR, Peters RM, Li J, Rao SD, Woodcroft KJ, Cassidy-Bushrow AE. Early pregnancy vitamin D and patterns of antenatal inflammation in African-American women. J Reprod Immunol. 2015 Feb;107:52-8. doi: 10.1016/j.jri.2014.09.054. Epub 2014 Oct 14. PMID 25453750
- [Background] Hypponen E, Cavadino A, Williams D, Fraser A, Vereczkey A, Fraser WD, Banhidy F, Lawlor D, Czeizel AE. Vitamin D and pre-eclampsia: original data, systematic review and meta-analysis. Ann Nutr Metab. 2013;63(4):331-40. doi: 10.1159/000358338. Epub 2014 Feb 28. PMID 24603503
- [Background] Theodoratou E, Tzoulaki I, Zgaga L, Ioannidis JP. Vitamin D and multiple health outcomes: umbrella review of systematic reviews and meta-analyses of observational studies and randomised trials. BMJ. 2014 Apr 1;348:g2035. doi: 10.1136/bmj.g2035. PMID 24690624
- [Background] Bodnar LM, Platt RW, Simhan HN. Early-pregnancy vitamin D deficiency and risk of preterm birth subtypes. Obstet Gynecol. 2015 Feb;125(2):439-447. doi: 10.1097/AOG.0000000000000621. PMID 25569002
- [Background] Liu PT, Stenger S, Li H, Wenzel L, Tan BH, Krutzik SR, Ochoa MT, Schauber J, Wu K, Meinken C, Kamen DL, Wagner M, Bals R, Steinmeyer A, Zugel U, Gallo RL, Eisenberg D, Hewison M, Hollis BW, Adams JS, Bloom BR, Modlin RL. Toll-like receptor triggering of a vitamin D-mediated human antimicrobial response. Science. 2006 Mar 24;311(5768):1770-3. doi: 10.1126/science.1123933. Epub 2006 Feb 23. PMID 16497887
- [Background] Thota C, Farmer T, Garfield RE, Menon R, Al-Hendy A. Vitamin D elicits anti-inflammatory response, inhibits contractile-associated proteins, and modulates Toll-like receptors in human myometrial cells. Reprod Sci. 2013 Apr;20(4):463-75. doi: 10.1177/1933719112459225. Epub 2012 Sep 25. PMID 23012315
- [Background] Arora CP & Hobel, C. Vitamin D - a novel role in pregnancy. Bioploymers and Cell. 2010;26(97):104.
- [Background] Accortt EE, Schetter CD, Peters RM, Cassidy-Bushrow AE. Lower prenatal vitamin D status and postpartum depressive symptomatology in African American women: Preliminary evidence for moderation by inflammatory cytokines. Arch Womens Ment Health. 2016 Apr;19(2):373-83. doi: 10.1007/s00737-015-0585-1. Epub 2015 Sep 26. PMID 26407996
- [Background] Parcells DA. Women's mental health nursing: depression, anxiety and stress during pregnancy. J Psychiatr Ment Health Nurs. 2010 Nov;17(9):813-20. doi: 10.1111/j.1365-2850.2010.01588.x. PMID 21040227
- [Background] Burt VK, Stein K. Epidemiology of depression throughout the female life cycle. J Clin Psychiatry. 2002;63 Suppl 7:9-15. PMID 11995779
- [Background] Davalos DB, Yadon CA, Tregellas HC. Untreated prenatal maternal depression and the potential risks to offspring: a review. Arch Womens Ment Health. 2012 Feb;15(1):1-14. doi: 10.1007/s00737-011-0251-1. Epub 2012 Jan 4. PMID 22215285
- [Background] Grote NK, Bridge JA, Gavin AR, Melville JL, Iyengar S, Katon WJ. A meta-analysis of depression during pregnancy and the risk of preterm birth, low birth weight, and intrauterine growth restriction. Arch Gen Psychiatry. 2010 Oct;67(10):1012-24. doi: 10.1001/archgenpsychiatry.2010.111. PMID 20921117
- [Background] Szegda K, Markenson G, Bertone-Johnson ER, Chasan-Taber L. Depression during pregnancy: a risk factor for adverse neonatal outcomes? A critical review of the literature. J Matern Fetal Neonatal Med. 2014 Jun;27(9):960-7. doi: 10.3109/14767058.2013.845157. Epub 2013 Oct 17. PMID 24044422
- [Background] Accortt EE, Cheadle AC, Dunkel Schetter C. Prenatal depression and adverse birth outcomes: an updated systematic review. Matern Child Health J. 2015 Jun;19(6):1306-37. doi: 10.1007/s10995-014-1637-2. PMID 25452215
- [Background] Hu R, Li Y, Zhang Z, Yan W. Antenatal depressive symptoms and the risk of preeclampsia or operative deliveries: a meta-analysis. PLoS One. 2015 Mar 19;10(3):e0119018. doi: 10.1371/journal.pone.0119018. eCollection 2015. PMID 25789626
- [Background] Furuta M, Sandall J, Cooper D, Bick D. The relationship between severe maternal morbidity and psychological health symptoms at 6-8 weeks postpartum: a prospective cohort study in one English maternity unit. BMC Pregnancy Childbirth. 2014 Apr 7;14:133. doi: 10.1186/1471-2393-14-133. PMID 24708797
- [Background] Goodman JH. Postpartum depression beyond the early postpartum period. J Obstet Gynecol Neonatal Nurs. 2004 Jul-Aug;33(4):410-20. doi: 10.1177/0884217504266915. PMID 15346666
- [Background] Kendler KS, Neale MC, Kessler RC, Heath AC, Eaves LJ. The lifetime history of major depression in women. Reliability of diagnosis and heritability. Arch Gen Psychiatry. 1993 Nov;50(11):863-70. doi: 10.1001/archpsyc.1993.01820230054003. PMID 8215812
- [Background] Georgiopoulos AM, Bryan TL, Wollan P, Yawn BP. Routine screening for postpartum depression. J Fam Pract. 2001 Feb;50(2):117-22. PMID 11219558
- [Background] Bryan TL, Georgiopoulos AM, Harms RW, Huxsahl JE, Larson DR, Yawn BP. Incidence of postpartum depression in Olmsted County, Minnesota. A population-based, retrospective study. J Reprod Med. 1999 Apr;44(4):351-8. PMID 10319305
- [Background] Beck CT, Gable RK, Sakala C, Declercq ER. Posttraumatic stress disorder in new mothers: results from a two-stage U.S. national survey. Birth. 2011 Sep;38(3):216-27. doi: 10.1111/j.1523-536X.2011.00475.x. Epub 2011 May 20. PMID 21884230
- [Background] The American College of Obstetricians and Gynecologists Committee Opinion no. 630. Screening for perinatal depression. Obstet Gynecol. 2015 May;125(5):1268-1271. doi: 10.1097/01.AOG.0000465192.34779.dc. PMID 25932866
- [Background] Siu AL; US Preventive Services Task Force (USPSTF); Bibbins-Domingo K, Grossman DC, Baumann LC, Davidson KW, Ebell M, Garcia FA, Gillman M, Herzstein J, Kemper AR, Krist AH, Kurth AE, Owens DK, Phillips WR, Phipps MG, Pignone MP. Screening for Depression in Adults: US Preventive Services Task Force Recommendation Statement. JAMA. 2016 Jan 26;315(4):380-7. doi: 10.1001/jama.2015.18392. PMID 26813211
- [Background] Chaudron LH, Wisner KL. Perinatal depression screening: let's not throw the baby out with the bath water! J Psychosom Res. 2014 Jun;76(6):489-91. doi: 10.1016/j.jpsychores.2014.03.011. Epub 2014 Mar 28. No abstract available. PMID 24840147
- [Background] Thombs BD, Arthurs E, Coronado-Montoya S, Roseman M, Delisle VC, Leavens A, Levis B, Azoulay L, Smith C, Ciofani L, Coyne JC, Feeley N, Gilbody S, Schinazi J, Stewart DE, Zelkowitz P. Depression screening and patient outcomes in pregnancy or postpartum: a systematic review. J Psychosom Res. 2014 Jun;76(6):433-46. doi: 10.1016/j.jpsychores.2014.01.006. Epub 2014 Jan 28. PMID 24840137
- [Background] Le Strat Y, Dubertret C, Le Foll B. Prevalence and correlates of major depressive episode in pregnant and postpartum women in the United States. J Affect Disord. 2011 Dec;135(1-3):128-38. doi: 10.1016/j.jad.2011.07.004. Epub 2011 Jul 29. PMID 21802737
- [Background] Austin MP; Marce Society Position Statement Advisory Committee. Marce International Society position statement on psychosocial assessment and depression screening in perinatal women. Best Pract Res Clin Obstet Gynaecol. 2014 Jan;28(1):179-87. doi: 10.1016/j.bpobgyn.2013.08.016. Epub 2013 Sep 3. PMID 24138943
- [Background] Wells KB, Sherbourne C, Schoenbaum M, Duan N, Meredith L, Unutzer J, Miranda J, Carney MF, Rubenstein LV. Impact of disseminating quality improvement programs for depression in managed primary care: a randomized controlled trial. JAMA. 2000 Jan 12;283(2):212-20. doi: 10.1001/jama.283.2.212. PMID 10634337
- [Background] Kingston DE, Biringer A, McDonald SW, Heaman MI, Lasiuk GC, Hegadoren KM, McDonald SD, Veldhuyzen van Zanten S, Sword W, Kingston JJ, Jarema KM, Vermeyden L, Austin MP. Preferences for Mental Health Screening Among Pregnant Women: A Cross-Sectional Study. Am J Prev Med. 2015 Oct;49(4):e35-43. doi: 10.1016/j.amepre.2015.03.026. Epub 2015 Jul 3. PMID 26143952
- [Background] Segre LS, Orengo-Aguayo RE, Siewert RC. Depression Management by NICU Nurses: Mothers' Views. Clin Nurs Res. 2016 Jun;25(3):273-90. doi: 10.1177/1054773815592596. Epub 2015 Jul 2. PMID 26137943
- [Background] Feeley N, Bell L, Hayton B, Zelkowitz P, Carrier ME. Care for Postpartum Depression: What Do Women and Their Partners Prefer? Perspect Psychiatr Care. 2016 Apr;52(2):120-30. doi: 10.1111/ppc.12107. Epub 2015 Feb 25. PMID 25711930
- [Background] Venkatesh KK, Riley L, Castro VM, Perlis RH, Kaimal AJ. Association of Antenatal Depression Symptoms and Antidepressant Treatment With Preterm Birth. Obstet Gynecol. 2016 May;127(5):926-933. doi: 10.1097/AOG.0000000000001397. PMID 27054941
- [Background] Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 report on dietary reference intakes for calcium and vitamin D from the Institute of Medicine: what clinicians need to know. J Clin Endocrinol Metab. 2011 Jan;96(1):53-8. doi: 10.1210/jc.2010-2704. Epub 2010 Nov 29. PMID 21118827
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Horowitz M, Wilner N, Alvarez W. Impact of Event Scale: a measure of subjective stress. Psychosom Med. 1979 May;41(3):209-18. doi: 10.1097/00006842-197905000-00004. PMID 472086
- [Background] Cohen S. Perceived stress in a probability sample of the United States. Sage Publications, Inc. 1988:31-67.
- [Background] Campbell-Sills L, Norman SB, Craske MG, Sullivan G, Lang AJ, Chavira DA, Bystritsky A, Sherbourne C, Roy-Byrne P, Stein MB. Validation of a brief measure of anxiety-related severity and impairment: the Overall Anxiety Severity and Impairment Scale (OASIS). J Affect Disord. 2009 Jan;112(1-3):92-101. doi: 10.1016/j.jad.2008.03.014. Epub 2008 May 16. PMID 18486238
- [Background] Spitzer RL, Williams JB, Gibbon M, First MB. The Structured Clinical Interview for DSM-III-R (SCID). I: History, rationale, and description. Arch Gen Psychiatry. 1992 Aug;49(8):624-9. doi: 10.1001/archpsyc.1992.01820080032005. PMID 1637252
- [Background] Lobbestael J, Leurgans M, Arntz A. Inter-rater reliability of the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID I) and Axis II Disorders (SCID II). Clin Psychol Psychother. 2011 Jan-Feb;18(1):75-9. doi: 10.1002/cpp.693. PMID 20309842
- [Background] Mossner R, Mikova O, Koutsilieri E, Saoud M, Ehlis AC, Muller N, Fallgatter AJ, Riederer P. Consensus paper of the WFSBP Task Force on Biological Markers: biological markers in depression. World J Biol Psychiatry. 2007;8(3):141-74. doi: 10.1080/15622970701263303. PMID 17654407
- [Background] Gemmill AW, Leigh B, Ericksen J, Milgrom J. A survey of the clinical acceptability of screening for postnatal depression in depressed and non-depressed women. BMC Public Health. 2006 Aug 17;6:211. doi: 10.1186/1471-2458-6-211. PMID 16914061
- See also: Maternal Mental Health NOW Referral Directory — http://directory.maternalmentalhealthnow.org/